CLINICAL TRIAL: NCT05493319
Title: Effects of Hypopressive Exercise Associated With Strength and Resistance Training in the Management of Fatigue, Urinary Incontinence Symptoms, Sexual Function and Quality of Life in Women Treated for Gynecological Cancer
Brief Title: Hypopressive Exercise Associated With Strength and Resistance Training in Women Treated for Gynecological Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Ivana Leão Ribeiro, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCM
Record Dates: First submitted 2022-07-09; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Gynecologic Cancer
Keywords: Exercise Therapy; Neoplasms; Fatigue; Quality of Life; Urinary Incontinence
MeSH Terms: conditions — Neoplasms; Fatigue; Urinary Incontinence | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-blind randomized clinical trial: interventional group and usual care group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments before and after the intervention will be performed by a physical therapist blinded to the allocation of participants in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypopresive, strength and resistance exercises (Experimental): Participants will perform 3 types of hypopresive exercises in the end of strength and resistance exercises intervention.
  Interventions: Other: Exercises
- Strength and resistance exercises (Active Comparator): Participants will perform strength and resistance exercises intervention.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Both groups will train three times a week, twice synchronously online and once asynchronously, considering a standardized exercise guideline. In all intervention sessions, conventional exercises will be guided by the standardized exercise guideline previously developed by the study team, for 4 weeks. Hypopresive, strength and resistance exercises group will receive static hypopressive exercise in supine position, with variant of arms in flexion, abduction and extension, consisting of 3 exercises at the end of the intervention with strength and resistance exercises.

SUMMARY:
The study aims to evaluate the effects of 4 weeks of hypopressive exercise associated with resistance training and aerobic exercises on fatigue, symptoms of urinary incontinence, sexual function and quality of life in women treated for gynecological cancer compared to a group that will perform conventional training. .

DETAILED DESCRIPTION:
Objective: To evaluate the effects of 4 weeks of hypopressive exercise associated with resistance training and aerobic exercises on fatigue, symptoms of urinary incontinence, sexual function and quality of life in women treated for gynecological cancer compared to a group that will perform conventional training.

Methods: This will be a single-blind randomized clinical trial. A hypopressive exercise intervention associated with resistance training and aerobic exercise will be carried out during twelve telerehabilitation sessions. Patients over 18 years of age who are diagnosed with gynecological cancer and who are indicated for radiotherapy or chemotherapy will participate. Patients will be randomly assigned to an experimental group of hypopressive exercises associated with resistance training and aerobic exercises or conventional training. Fatigue, quality of life, symptoms of urinary incontinence and sexual function will be evaluated before and after the intervention.

Discussion: The results of this clinical trial will determine the impact of conventional training associated with hypopressive exercise on the negative side effects of cancer treatment in women with gynecological cancer.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must have a medical diagnosis of gynecological cancer
* Participants should have an indication for chemotherapy or radiotherapy, associated or not with pelvic lymphadenectomy
* Women with an age range over 18 years with a limit of up to 60 years
* Participants who are able to practice physical activity

Exclusion Criteria:

* Recurrence of gynecological cancer
* Presence of lymphedema in the lower limb, measured by cytometry of the lower limb with a tape measure; asymmetries of more than 2 cm between the limbs were considered edema
* Diagnosis of metastasis
* Heart disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at 4 weeks in quality of life assessed by a questionnaire | Baseline/up to 4 weeks
  Data are be collected using the questionnaire The European Organization for Research and Treatment of Cancer Core Quality of Life questionnaire it contains 30 items and the total score ranges from 0 (very poor) to 100 (excellent) for the functional dimensions, and from 0 (excellent) to 100 (very poor) for the symptom dimensions. All of the multi-item scales and single-item measures range in a score from 0 to 100, where a high score represents a higher response level.
Change from baseline at 4 weeks in sexual function assessed by a questionnaire | Baseline/up to 4 weeks
  Data are be collected using the questionnaire Organ Prolapse/Urinary Incontinence Sexual Questionnaire that consists of 12 items, the scores range from 0 to 48, the higher the score, the better the sexual function.
Change from baseline at 4 weeks in urinary incontinence assessed by a questionnaire | Baseline/up to 4 weeks
  Data are be collected using the questionnaire Pelvic Floor Impact Questionnaire-Short Form 7 that score corresponds to 0: not at all; 1: something; 2: moderately and 3: quite a bit. For the conversion of the score, the mean score must be multiplied with 100/3 and a scale range of 0 to 100 is obtained, the higher the score, the greater the impact of symptoms on general activities.
Change from baseline at 4 weeks in fatigue assessed by a scale | Baseline/up to 4 weeks
  Data are be collected using the scale the Brief Fatigue Inventory that it is made up of 3 items, the categorization of fatigue levels can be obtained through an arithmetic average of the scores obtained in each item. Score 0 means "no fatigue"; 1-3: "mild fatigue"; 4-6: "moderate fatigue" and 7-10: "severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana L Ribeiro, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Catholic University of Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT05493319/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT05493319/ICF_001.pdf